CLINICAL TRIAL: NCT05576493
Title: Combined Phacoemulsification and Different Modes of Diode Laser Therapy in Management of Chronic Angle Closure Glaucoma. A Comparative Study
Brief Title: Combined Phacoemulsification and Diode Laser Therapy in Chronic Angle Closure Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fayrouz Aboalazayem, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-68-2022
Record Dates: First submitted 2022-10-08; First posted 2022-10-12 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Angle Closure Glaucoma
Keywords: angle closure glaucoma; cyclophotocoagulation
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A:phaco+MP-TSCPC (Experimental): 22 patients with primary angle closure glaucoma will undergo phacoemulsification and micropulse cyclophotocoagulation
  Interventions: Procedure: phaco+MP-TSCPC
- B:phaco+TSCPC (Experimental): 22 patients with primary angle closure glaucoma will undergo phaco and transscleral cyclophotocoagulation
  Interventions: Procedure: phaco+TSCPC
- C:phaco+endocyclophotocoagulation (Experimental): 22 patients with primary angle closure glaucoma will undergo phaco and endocyclophotocoagulation after cataract removal
  Interventions: Procedure: phaco+endocyclophotocoagulation
- D:phaco GSL (Experimental): 22 patients with primary angle closure glaucoma will undergo phaco and goniosynechiolysis
  Interventions: Procedure: phaco GSL

INTERVENTIONS:
Procedure: phaco+MP-TSCPC — The procedure starts with performing the cyclophotocoagulation using the Micropulse P3 device (IQ 810 Laser Systems; Iridex, Mountain View, CA, USA) at 2500 mW with a duration of 90 seconds in each hemisphere at a 31.3% duty cycle under local anesthesia and then performing phacoemulsification and IOL implantation.
  Arms: A:phaco+MP-TSCPC
Procedure: phaco+TSCPC — The procedure starts with performing the cyclophotocoagulation using the IRIDEX's G probe device (IRIDEX Corp. Mountain View, CA, USA) at 1500 to2000 mW with a duration of 1500 ms applying about 15 shots in one hemisphere only under local anesthesia and then performing phacoemulsification and IOL implantation.
  Arms: B:phaco+TSCPC
Procedure: phaco+endocyclophotocoagulation — phacoemulsification will be done and endocyclophotocoagulation will be done after cataract extraction
  Arms: C:phaco+endocyclophotocoagulation
Procedure: phaco GSL — phacoemulsification will be done and then the angle is visualized by direct goniolens then the synechia are dissected by cohesive viscoelastic.
  Arms: D:phaco GSL

SUMMARY:
comparing different types of cuclophotocoagulation with cataract extraction to cataract extraction and goniocynechiolysis in cases of chronic angle closure glaucoma

DETAILED DESCRIPTION:
Evaluation of the safety of MP-TSCPC , CW-TSCPC and endoscopic cyclophotocoagulation when combined with phacoemulsification in cases with CACG Comparing the efficacy of the combined procedures in control of the IOP and the success rate versus lens extraction combined with synechiolysis

ELIGIBILITY:
Inclusion Criteria:

* Patients between 20 to 70 years

chronic angle closure glaucoma

Exclusion Criteria:

* Patients in acute attack of angle closure.
* Patients with previous filtering surgery or cycloablative procedure

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
the percentage of intraocular pressure change | 6 Months
  measuring the intraocular pressure after 1M, 3M and 6M

SECONDARY OUTCOMES:
percent change of antiglaucoma medications | 6 Months
  the number of medication before and after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelrahman, PhD, Study Chair — kasr alainy
Locations (1):
- Kasr Alainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No